CLINICAL TRIAL: NCT06933303
Title: Distraction as Treatment for Pain in Children in Resource-scarce Settings
Acronym: DISTRACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vrinnevi Hospital (Other)
Collaborators: Radboud University Medical Center (Other); Linkoeping University (Other Government); University of KwaZulu (Other)
Responsible Party: Principal Investigator, Måns Muhrbeck MD, PhD, Principal investigator, Vrinnevi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DISTRACT-01
Record Dates: First submitted 2025-04-08; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Pain, Acute
Keywords: Distraction; Pain; Burn injury; Dressing change; Pediatric
MeSH Terms: conditions — Acute Pain; Pain; Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Undergoing dressing change with standard medical care. Standard medical care can include: no pain alleviation methods; paracetamol; non-steroidal anti-inflammatory drug; combination of paracetamol with non-steroidal anti-inflammatory drug
- Distraction (Experimental): Undergoing dressing change with standard medical care (as described above for Control arm), combined with distraction by use of a kaleidoscope as a possible pain alleviation method.
  Interventions: Device: Distraction with kaleidoscope

INTERVENTIONS:
Device: Distraction with kaleidoscope — During the intervention measurement, the pediatric patient will be distracted by the use of a kaleidoscope during the procedure. Distraction by use of the kaleidoscope will be initiated at the start of the procedure (dressing change) and the kaleidoscope will be offered until at least a minute after the procedure is completed. Removal of the dressing will be started when the child seems distracted as indicated by response with a smile or laughter, or a verbal response
  Arms: Distraction

SUMMARY:
Pain alleviation in pediatric patients can be challenging for medical professionals working in resource scarce settings due to limited availability of medication, monitoring equipment, or training in this field of expertise. This poses the need for a readily available tool for pain reduction that does not rely on expensive equipment or medication and which can easily be applied in resource scarce settings around the world. With this research project we aim to assess the effectiveness of a simple, inexpensive, non-electronic distraction method: a kaleidoscope, to reduce acute pain in pediatric patients undergoing dressing changes in resource scarce environments.

A randomized controlled trial will be performed at the Edendale Hospital in Pietermaritzburg KwaZulu Natal, South Africa. Pediatric patients between the age of 7-12 years with partial thickness burn injuries who require dressing changes in the outpatient clinic will be randomized into two groups: one group (control) will receive standard practice of care which concerns a dressing change without any pain alleviation other than paracetamol or a non-steroidal anti inflammatory drug (NSAID), and one group (intervention) will receive distraction by use of a kaleidoscope as method for potential pain alleviation on top of standard medical care. The primary outcome will be the difference in mean change in pain score (from before to during the dressing change) between the control and distraction group.

This study is expected to demonstrate that the use of a non-electronic distraction technique effectively alleviates pain in children undergoing dressing changes and that its use is feasible in low resource settings. The distraction technique can be applied as add-on to pharmacological treatment, or stand-alone when no pharmacological treatment is available. Distraction is expected to be safe and can even be applied by an accompanying parent, resulting in lower barriers for healthcare workers to apply it. Appropriate pain relief will improve psychological wellbeing of pediatric patients undergoing painful procedures, and it might even improve recovery and physical rehabilitation since pain has been associated with physical as well as mental morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients between the age of 7 and 12 years old with burn injuries requiring dressing changes in the outpatient clinic, who in regular practice (non-research setting) would not receive any analgesics;
* Type of burn injury: partial thickness burns with a burned area not greater than 10% at the moment of the first dressing change measurement as part of this research

Exclusion Criteria:

* Patients who received split skin grafts for their burns;
* Patients on sedatives or anti-epileptics;
* The use of pain-relieving medication other than paracetamol or ibuprofen;
* Painful additional injuries other than the burn injury;
* Patients who are nursed in isolation;
* Physical or mental impairments which make it impossible to adequately comply with the trial protocol. For example, visual impairments, impaired ability to communicate, psychological comorbidities, and burns that limit the use of a kaleidoscope (facial burns or burns to both hands);
* Retrospective exclusion if the patient in the intervention group did not look through the kaleidoscope for more than 50% of the procedure time.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 126 (Estimated)
Dates: Start 2025-03-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in pain score | Pain scores measured five minutes prior to dressing change; pain score during dressing change, measured immediately after removal of the dressing
  The change (increase) in pain scores (the Wong-Baker FACES Pain Rating Scale and the FLACC scale), 0 (less pain)-10 (more pain) , from prior to the dressing change to during the dressing change

SECONDARY OUTCOMES:
Postprocedural pain score decrease | Pain scores during dressing change, after removal of the dressing; pain score at five minutes after dressing change
  Change in mean pain scores (the Wong-Baker FACES Pain Rating Scale and the FLACC scale), 0 (less pain)-10 (more pain) , when comparing scores during with scores after the procedure.
Heart rate | Measured five minutes before dressing change; measured during dressing change at two-minute interval; measured five minutes after dressing change
  Change/course of heart rate before, during and after dressing change
Oxygen saturation | Measured five minutes before dressing change; measured during dressing change at two-minute interval; measured five minutes after dressing change
  Change/course of blood oxygen levels before, during and after dressing change
Global satisfaction | Five minutes after dressing change
  Global judgement of satisfaction with treatment by caregiver and medical professional, will be measured on a 1 (very dissatisfied)-5 (very satisfied) scale based on the question: "Considering pain relief, side effects, and emotional status, how satisfied were you with the dressing change the child underwent?"
Procedure time | Duration of dressing change
  Procedure time (seconds), reflecting procedure efficiency/patient cooperation

CONTACTS AND LOCATIONS:
Locations (1):
- Ngwelezana Hospital, Empangeni, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: No